CLINICAL TRIAL: NCT04878588
Title: The Correlation Between High Resolution Impedance Manometry and Videofluoroscopic Measurements of Swallowing Function After Patients Undergoing Esophagectomy
Brief Title: The Correlation Between the Barium Examination and High Resolution Impedance Manometry
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202102001RIND
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: the Correlation Between the Barium Examination and High Resolution Impedance Manometry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients receiving esophagectomy: the patients receiving esophagectomy during perioperative period. They receive barium examination and high resolution impedance manometry at the same time
  Interventions: Other: patients received high resolution impedance manometry

INTERVENTIONS:
Other: patients received high resolution impedance manometry — patients received the above two examination at the same time
  Other Names: patients received barium examination

SUMMARY:
In many cases, the manometric examination is not feasible because of the pharyngeal sinusitis or pharyngeal torsion. In addition, although previous conventional manometry was used to estimate pharyngeal swallowing, the bolus flow transmission was still not evaluated, which still depended on the videofluoscopic swallowing studies. High resolution impedance manometry could help us to measure the bolus flow according to the impedance changes. However, the comparison between two approach methods of postoperative recovery of swallowing function is still inconclusive. In this study, we aimed to examine the correlation between high-resolution manometric and videofluoroscopic (Barium) measurements of the swallowing function.

DETAILED DESCRIPTION:
In many cases, the manometric examination is not feasible because of the pharyngeal sinusitis or pharyngeal torsion. In addition, although previous conventional manometry was used to estimate pharyngeal swallowing, the bolus flow transmission was still not evaluated, which still depended on the videofluoscopic swallowing studies. High resolution impedance manometry (HRIM) could help us to measure the bolus flow according to the impedance changes. However, the comparison between two approach methods of postoperative recovery of swallowing function is still inconclusive.

In this study, we aimed to examine the correlation between high-resolution manometric and videofluoroscopic (Barium) measurements of the swallowing function.

For the patients and method decription, consecutive patients who will fulfill the criteria of elective esophagectomy patients aged >= 20 will be enrolled. After got the inform consent, these patients receive the swallowing function by barium examination and HRIM.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving elective esopagectomy

Exclusion Criteria:

* patients with major organ disease, such as heart, lung, or liver disease
* patients with coagulopathy

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients receiving elective esophagectomy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-09-06 (Estimated); Primary Completion 2025-05-10 (Estimated); Study Completion 2027-05-10 (Estimated)

PRIMARY OUTCOMES:
the contractility of the muscle at the upper gastrointestinal tract | 20 minutes
  the contractility at the upper gastrointestinal tract muscle

IPD SHARING:
Plan to Share IPD: No
due to ethical issue